CLINICAL TRIAL: NCT04884048
Title: Multicentric Study for the Validation and Improvement of a Structured Report Tool for the Imaging Characterization of Bone Tumors - Bone Tumor Imaging Report and Data System (BTI-RADS)
Brief Title: Multicentric Bone Tumor Imaging Report and Data System
Acronym: BTI-RADS M
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Groupement des Hopitaux de l'institut catholique de Lille (Unknown); Hôpital Cochin (Other); Hopital Jules Courmont - Centre Hospitalier Lyon Sud (Other); Centre Hospitalier Universitaire de Besancon (Other); Centre Oscar Lambret (Other); Hospital Purpan (Other); University Hospital, Lille (Other); University Hospital, Bordeaux (Other)
Responsible Party: Principal Investigator, Pedro TEIXEIRA-GONDIM, MD, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: CentralHNF BTI-RADSM
Record Dates: First submitted 2021-05-07; First posted 2021-05-12 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Bone Neoplasm
Keywords: Bone Neoplasms; Multidetector Computed Tomography; Radiographs; Magnetic Resonance Imaging; Evidence-Based Medicine
MeSH Terms: conditions — Bone Neoplasms | interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Benign bone tumors: Patients with benign lesions confirmed either by histology or imaging follow-up showing lesion stability.
  Interventions: Diagnostic Test: Radiographs
- Malignant bone tumors: Patients with malignant lesions confirmed by histology.
  Interventions: Diagnostic Test: Radiographs

INTERVENTIONS:
Diagnostic Test: Radiographs — Analysis of the images acquired for the initial characterization of bone lesions using a systematic report system
  Other Names: CT; MRI

SUMMARY:
In this study a previously described structured multimodality image report system for the characterization of focal bone lesions is evaluated in a larger patient population. The objective of this study is to evaluate the performance of this tool stratifying the malignancy risk of bone tumors.

DETAILED DESCRIPTION:
The characterization of focal bone lesions by imaging can be difficult. Primary bone sarcomas are rare, accounting for 0.2% of all malignant tumors occurring at an estimated rate of one tenth that of soft tissue sarcomas. Focal bone lesions have a wide differential diagnosis, including benign and malignant neoplasms, metabolic disorders, degenerative changes, and tumor-like conditions. The precise differentiation between benign and malignant bone tumors is essential for optimal patient management, with a considerable impact on prognosis and survival rates. The relapse-free survival of patients with sarcoma is significantly better when treatment is guided by a multidisciplinary oncology committee. In addition, surgical treatment in referral centers reduces the risk of recurrence and death.

Due to the rarity of primary malignant bone neoplasms and the varied imaging presentation of focal bone lesions, radiologists outside of cancer centers tend to have little experience with this type of abnormality. Thus, imaging reports can be unclear and misleading, increasing the risk of misdiagnosis and suboptimal patient management. Previous studies have largely addressed the specific imaging features of bone tumors, and a systematic approach to the assessment of bone tumors has been recommended. However, there is little information on how to combine these imaging results and which are most relevant for characterization of lesions.

Various studies have demonstrated the value of structured analysis of medical information in clinical decision making and such an approach is currently used for the assessment of malignancy in various organs and systems. For bone tumors, this approach requires the combined analysis of several demographic, clinical and imaging characteristics. Of the large number of features described, 16 (seven benign and nine malignant) were considered relevant for the differentiation between benign and malignant tumors. Three signs (Lodwick-Madewell grade III, aggressive periosteal reaction and suspected or confirmed metastatic disease) had a mean frequency of associated malignancy greater than 80%. Thus, lesions showing any of these signs should be considered malignant until proven otherwise. It should be noted that these 3 signs are CT or standard radiography criteria, confirming the essential role of X-ray-based methods for the characterization of bone tumors. On the contrary, certain signs classically suggestive of malignancy, such as a history of pain, pathological fracture and endosteal scalloping, have been identified as non-determining indicators for the characterization of these lesions. These data could contribute to a more precise assessment of the aggressive potential of a bone tumor. Finally, on the basis of these results, an evidence-based classification of solitary bone lesions (BTI-RADS) was proposed, allowing the stratification of bone tumors into four classes with an average frequency of malignancy of 0%; 2.2% (1.1 - 3.1%), 20.1% (17 - 24.4%) and 71% (65.6 - 75%) for each class. This system was applicable for readers with different levels of expertise, including a general radiologist, with acceptable interobserver reproducibility (Kappa = 0.67). BTI-RADS could be particularly beneficial outside of specialized oncology centers.

However, the BTI-RADS was established based on a single-center analysis of a relatively small patient population. The application of this system in a larger population in multicentric study is necessary to validate this tool and potentially refine it through the identification of additional pertinent criteria for lesion characterization.

ELIGIBILITY:
Inclusion Criteria:

* Patient evaluated for the initial imaging characterization of a focal bone lesion.
* Availability of conventional radiographs or a CT study for patients with lesions in the spine, pelvis or calvarium.
* Availability of a contrast enhanced MRI study.

Exclusion Criteria:

* Prio surgery
* History of neoadjuvant threatment
* Contra-indications to contrast enhanced MRI
* Diffuse bone pathology

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients referred for the initial imaging characterization of focal bone lesions.
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Structured report item analysis | 30 minutes
  Each component of the structure report system will be analyzed and compared between the study groups.

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - University hospital of Nancy, Nancy, Grand Est
  - Hôpital Universitaire Paris Centre site Cochin APHP, Paris, Ille de France
  - Centre Oscar Lambret, Lille, Nord
  - Groupement des Hopitaux de l'institut catholique de Lille, Lille, Nord
  - CHRU Lille, Lille, Nord
  - CHRU Besançon, Besançon
  - Chu Bordeaux, Bordeaux
  - Université Lyon 1 - Centre Hospitalier Lyon-Sud, Lyon
  - Hôpital de Purpan - CHU Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ribeiro GJ, Gillet R, Hossu G, Trinh JM, Euxibie E, Sirveaux F, Blum A, Teixeira PAG. Solitary bone tumor imaging reporting and data system (BTI-RADS): initial assessment of a systematic imaging evaluation and comprehensive reporting method. Eur Radiol. 2021 Oct;31(10):7637-7652. doi: 10.1007/s00330-021-07745-9. Epub 2021 Mar 25. PMID 33765161